CLINICAL TRIAL: NCT02675010
Title: Value of Additional Corpus Biopsy for Diagnosis of H Pylori in Atrophic Gastritis. Prospective Non-randomized Multicenter Study
Brief Title: Value of Additional Corpus Biopsy for Diagnosis of H Pylori in Atrophic Gastritis. Prospective Non-randomized Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, MOHAMED ABDELLATIF, ass. prof., Mansoura University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: H1
Record Dates: First submitted 2016-02-02; First posted 2016-02-05 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2016-02

CONDITIONS: Helicobacter Pylori; Gastric Antrum; CORPUS BIOPSIES

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ENDOSCOPIC GASTRIC BIOPSIES (Other): ENDOSCOPIC BIOPSEIS TAKEN FROM BOTH ANTRUM AND CORPUS FOR H PYLORI DETECTION
  Interventions: Other: ENDOSCOPIC GASTRIC BIOPSIES FROM ANTRUM AND BODY

INTERVENTIONS:
Other: ENDOSCOPIC GASTRIC BIOPSIES FROM ANTRUM AND BODY — ENDOSCOPIC GASTRIC BIOPSIES FROM ANTRUM AND BODY

SUMMARY:
There are controversies about the best sites -biopsy based -tests for H pylori associated gastritis. The study is designed to evaluate the optimal site of gastric mucosal biopsy for identification of Helicobacter pylori, especially in case of gastric atrophy and/or intestinal metaplasia.

DETAILED DESCRIPTION:
. The study is designed to evaluate the optimal site of gastric mucosal biopsy for identification of Helicobacter pylori, especially in case of gastric atrophy and/or intestinal metaplasia. 400 patients with dyspepsia are planned to be enrolled in this study. in addition to the routine antral biospy, corpus biospies are taken to evaluate the optimal site of gastric mucosal biopsy for identification of Helicobacter pylori, especially in case of gastric atrophy and/or intestinal metaplasia.

ELIGIBILITY:
Inclusion Criteria:

* Patients included in this study are those with peptic ulcer disease, previous upper gastrointestinal surgery, a known or a suspected past history of H.pylori eradication therapy, a personal or first-degree family history of gastric cancer

Exclusion Criteria:

* those having received antibiotic or proton pump inhibitor treatment one month beforehand

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2014-06; Primary Completion 2016-06 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
H PYLORI POSITIVITY | 2 YEARS

CONTACTS AND LOCATIONS:
Overall Officials: MOHAMED ABDELLATIF, ASS PROF, Study Chair — MANSOURA FACULTY OF MEDICINE
Locations (1):
- Mansoura University Hospital, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: Undecided